CLINICAL TRIAL: NCT00207480
Title: Brief, Behavioral Intervention to Reduce Douching Among Adolescent and Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Tulane University School of Public Health and Tropical Medicine (Other)
Allocation: Randomized | Masking: None | Purpose: Other
Other Study IDs: CDC-NCHSTP-4415; U36/CCU300430-24
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Vaginal Douching; Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Motivational Interviewing

INTERVENTIONS:
Behavioral: Brief, motivational interviewing intervention

SUMMARY:
This study will implement and test a brief, tailored individual-level intervention to be used in two New Orleans adolescent clinics with female patients aged 16-24 who douche.

DETAILED DESCRIPTION:
The study implements a client-centered behavioral intervention (CCBI) based on Prochaska's Transtheoretical Model of Change (TMC) and the intervention will use Miller's Motivational Interviewing (MI) techniques. This intervention will be evaluated using (1) an audio/computer-assisted self-administered interview (ACASI) survey to assess changes in respondents' douching knowledge, attitudes, and practices, and (2) biological testing for Bacterial Vaginosis.

ELIGIBILITY:
Inclusion Criteria:

* Women attending between the ages of 16 and 24 who have douched at least once in the last 180 days, agree to a test for Bacterial Vaginosis, and agree to allow us to contact you by telephone or in person for a follow-up interview and testing for bacterial vaginosis.

Exclusion Criteria:

* currently pregnant, non-English speaking

Ages: 16 Years to 24 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0
Dates: Start 2004-10; Primary Completion 2004-10 (Actual); Study Completion 2004-10

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Kissinger, PhD, RN, Principal Investigator — Tulane University School of Public Health and Tropical Medicine
Locations (1):
- Orleans Women's Health Clinic, New Orleans, Louisiana, United States